CLINICAL TRIAL: NCT05782231
Title: Addressing the Epidemic of Chronic Pain Among Older Adults in Underserved Communities; The GetActive+ Study
Brief Title: Improving Health for Older Adults With Pain Through Engagement (Open-pilot)
Acronym: iHOPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Ana-Maria Vranceanu, PhD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023P000362
Record Dates: First submitted 2023-02-23; First posted 2023-03-23 (Actual); Results first posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Chronic Pain; Musculoskeletal Pain
Keywords: Older adults; Mind-body intervention; Chronic pain; Community health center; Physical function
MeSH Terms: conditions — Chronic Pain; Musculoskeletal Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GetActive+ (Experimental): A mind-body program focused on increasing physical and emotional function in older adults with chronic musculoskeletal pain
  Interventions: Behavioral: GetActive+

INTERVENTIONS:
Behavioral: GetActive+ — 10-week group mind body program focused on improving self-report, performance-based and ambulatory step count by combining mind body skills tailored for individuals with chronic pain, with gradual increased in walking using quota-based pacing and goal setting, adapted specifically for older adults from a medically underserved location.

SUMMARY:
The goal of this project is to conduct an open-pilot (N=30) to evaluate the feasibility, acceptability, and fidelity of a mind-body and activity program (GetActive+) with older adults with chronic pain. The investigators will test for improvements in self-reported, performance-based (i.e., six-minute walk test), and objective (i.e., step-count) physical function, emotional function, as well as feasibility, acceptability and implementation markers. Participants will complete measures at baseline and post-intervention.

This study received support from and inclusion in the HEAL Initiative (https://heal.nih.gov/).

DETAILED DESCRIPTION:
The aim of this phase is to establish feasibility (primary), acceptability, and fidelity of GetActive+ and study procedures in an open pilot (N=30). Deliverables: GetActive+ will be feasible (≥75% agree to participate), acceptable (≥75% of those enrolled will complete 8/10 sessions) and delivered with fidelity (≥75% sessions delivered as intended).

Our patients will be older adults with chronic pain from Revere HealthCare Center.

The GetActive+ program will incorporate mind-body skills, cognitive behavioral and physical restoration skills (e.g., quota-based pacing) to help individuals increase self-reported, performance based and objective (step count) physical function. This program will teach participants four core skills: 1) weekly goal setting for gradual increase in time spent walking paired with activities of daily living that are meaningful and important to participants (i.e. walk instead of drive to the store; walk to the park with kids) 2) quota-based pacing (increasing walking goal gradually non-contingent of pain); 3) mind-body skills (e.g., diaphragmatic breathing to manage intense pain flares and pain anxiety; body scan to increase body awareness and reduce reactivity to pain sensations; mindfulness exercises to understand the transience of pain and change one's relationship with it; self-compassion when falling short of set goals); and 4) understand the downward spiral (e.g. how reducing activity perpetuates pain and disability), correct myths about pain or unhelpful pain-related thoughts that interfere with meeting program goals. Participants will be encouraged to complete their homework (logs for mind-body practice, physical activities) each day. Participants will be given the option to receive homework and session reminders via text messages from study staff. This between session contact will focus on increasing treatment adherence, maintaining engagement, and session reminders. The investigators will run groups primarily in English with an additional two groups in Spanish.

Baseline assessments and post-intervention assessments will include the six-minute walk test (6MWT), objective step count via ActiGraph, and self-reported measures including physical function, emotional function, pain, social support, and loneliness.

ELIGIBILITY:
Inclusion Criteria:

1. Older Adults (i.e., age >=55)
2. Diagnosed musculoskeletal chronic pain of any type (e.g., pain > 3 months)
3. Pain score >=4 (moderate) on the Numerical Rating Scale
4. Cognitively able to participate as measured by the Short Portable Mental Health questionnaires (e.g., <4 errors)
5. No self-reported current active, untreated psychotic or substance use disorder that would interfere with participation in the research study
6. Ability to complete the 6-minute walk test under supervision of study staff
7. Patient at Revere HealthCare Center who is cleared for participation by medical staff
8. English or Spanish fluency

Exclusion Criteria:

1. Current serious medical illness that is expected to worsen in the next 6 months (e.g., cancer)
2. Individuals who are unwilling or unable to wear the ActiGraph device

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2023-04-18 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2024-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ana-Maria Vranceanu, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Data can be accessed in the Vivli data repository
Supporting Information: Study Protocol, SAP
Time Frame: Data is currently available in the repository.
Access Criteria: No specialized tools will be needed to access the data other than what is noted on the Vivli website.
URL: https://doi.org/10.25934/PR00010109

REFERENCES:
- [Background] Greenberg J, Lin A, Popok PJ, Kulich RJ, Edwards RR, Vranceanu AM. Getting Active Mindfully: Rationale and Case Illustration of a Group Mind-body and Activity Program for Chronic Pain. J Clin Psychol Med Settings. 2021 Dec;28(4):706-719. doi: 10.1007/s10880-020-09758-w. Epub 2021 Jan 19. PMID 33469845
- [Background] Grunberg VA, Greenberg J, Mace RA, Bakhshaie J, Choi KW, Vranceanu AM. Fitbit Activity, Quota-Based Pacing, and Physical and Emotional Functioning Among Adults With Chronic Pain. J Pain. 2022 Nov;23(11):1933-1944. doi: 10.1016/j.jpain.2022.07.003. Epub 2022 Jul 29. PMID 35914640
- [Background] Popok PJ, Greenberg J, Gates MV, Vranceanu AM. A qualitative investigation of activity measurement and change following a mind-body activity program for chronic pain. Complement Ther Clin Pract. 2021 Aug;44:101410. doi: 10.1016/j.ctcp.2021.101410. Epub 2021 May 2. PMID 33971485
- [Background] McDermott K, Levey N, Brewer J, Ehmann M, Hooker JE, Pasinski R, Yousif N, Raju V, Gholston M, Greenberg J, Ritchie CS, Vranceanu AM. Improving Health for Older Adults With Pain Through Engagement: Protocol for Tailoring and Open Pilot Testing of a Mind-Body Activity Program Delivered Within Shared Medical Visits in an Underserved Community Clinic. JMIR Res Protoc. 2023 Dec 29;12:e52117. doi: 10.2196/52117. PMID 38157234
- Available data/document: Individual Participant Data Set: VIV0001019 — https://doi.org/10.25934/PR00010109

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was facilitated through posted Massachusetts General Hospital (MGH) Institutional Review Board-approved flyers in the clinic and the hospital's research recruitment site, and referrals from MGH Revere HealthCare Center physicians, nurses, psychologists, and other relevant staff.
Pre-assignment Details: All enrolled participants were assigned to the intervention, GetActive+.
Period: Overall Study
Arm/Group | GetActive+
Started | 33
Completed | 32
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | GetActive+
Number analyzed (Participants) | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.76 (8.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 3
  White | 14
  More than one race | 0
  Unknown or Not Reported | 14
Region of Enrollment [Number; unit: participants]
  United States | 33

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Intervention Completion
Description: >=75 of patients approached agree to participate in intervention
Time Frame: 10 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Experimental: GetActive+: A mind-body program focused on increasing physical and emotional function in older adults with chronic musculoskeletal pain
  GetActive+: This is a 10-week group mind body program focused on improving self- report, performance based and ambulatory step count by combining mind body skills tailored for individuals with chronic pain, with gradual increased in walking using quota based pacing and goal setting, adapted specifically for older adults from a medically underserved location.
Arm/Group | Experimental: GetActive+
Number analyzed (Participants) | 38
Participants | 33

2. Primary Outcome: Acceptability
Description: >=75% of enrolled participants complete at least 8/10 sessions
Time Frame: 10 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: GetActive+
Number analyzed (Participants) | 33
Participants | 31

3. Primary Outcome: Fidelity of Session Components, As Rated by Clinicians
Description: Clinician raters, with experience in intervention refinement or delivery, randomly selected 20% of all sessions to rate their components for this outcome. All sessions were audio-recorded. The overall number of units analyzed, which is reported below, refers to that 20% of the total number of sessions that were then analyzed for this outcome); the overall number of participants analyzed, which is also reported below, is the total number of participants in this study. Clinician raters used fidelity checklists to guide their ratings of the different session components. A session component was considered delivered as intended if the rater provided a score ≥8 (the scale was 1=poor to 10=outstanding). Reported here are the number of session components with a score ≥8, indicating successful delivery; the percentage of the total analyzed sessions that this represents is also calculated out below. The study benchmark we looked to meet for this fidelity measure was 75%.
Time Frame: Fidelity, as described above, was assessed periodically throughout the 11 months of the study, and is presented here as the sum total counts of all the high scoring components (again, described above) that were assessed over this 11 month time period.
Measure: Count of Units; unit: Number of session components
Units Other Than Participants: Number of session components
Arm/Group | Experimental: GetActive+
Number analyzed (Participants) | 33
Number analyzed (Number of session components) | 1170
Number of session components | 1145

4. Secondary Outcome: Physical Function - Performance-based
Description: 6-minute walk test (6MWT), assesses distance walked (in meters) in 6 minutes.
Time Frame: Baseline (0 weeks), Post-test (1 week after intervention completion)
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Experimental: GetActive+
Number analyzed (Participants) | 33
meters
  Baseline | 243.1 (82.6)
  Post-test | 277.0 (77.8)

5. Secondary Outcome: Physical Function - Objective
Description: Average step count with ActiGraph GT3X-BTLE
Time Frame: Baseline (0 weeks), Post-test (1 week after intervention completion)
Measure: Mean (Standard Deviation); unit: steps
Arm/Group | Experimental: GetActive+
Number analyzed (Participants) | 33
steps
  Baseline | 2561.4 (2013.4)
  Post-test | 2560.3 (1797.7)

6. Secondary Outcome: Short Form Brief Pain Inventory (BPI) Pain Severity and Interference Subscales
Description: The Short Form Brief Pain Inventory (BPI) pain severity subscale assesses pain at its worst, least, average, and current. Minimum = 0, maximum = 10. Higher scores indicate worse outcome. The interference subscale assesses pain interference in the last 24 hours. Minimum = 0, maximum = 10. Higher scores indicate worse interference.
Time Frame: Baseline (0 weeks), Post-test (1 week after intervention completion)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental: GetActive+
Number analyzed (Participants) | 33
units on a scale
  Baseline | 5.7 (1.8)
  Post-test | 4.4 (2.3)

7. Secondary Outcome: Patient Health Questionnaire-8 (PHQ-8)
Description: The Patient Health Questionnaire (PHQ-8) is an assessment of depressive symptoms. Total summary score with Minimum = 0, Maximum = 24. Higher scores indicate worse outcome.
Time Frame: Baseline (0 weeks), Post-test (1 week after intervention completion)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental: GetActive+
Number analyzed (Participants) | 33
units on a scale
  Baseline | 8.4 (6.0)
  Post-test | 5.7 (6.1)

8. Secondary Outcome: Generalized Anxiety Disorder Scale-7 (GAD-7);
Description: The Generalized Anxiety Disorder scale-7 (GAD-7) is an assessment of generalized anxiety symptoms. GAD-7 total score is obtained by adding the score for each of the items. Minimum = 0, Maximum = 21. Scores of 5-9 (mild), 10-14 (moderate), and 15-21 (severe) represent thresholds for mild, moderate, and severe anxiety. Higher scores indicate worse outcome.
Time Frame: Baseline (0 weeks), Post-test (1 week after intervention completion)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental: GetActive+
Number analyzed (Participants) | 33
units on a scale
  Baseline | 6.2 (5.4)
  Post-test | 5.1 (4.2)

9. Secondary Outcome: PROMIS Physical Function - Short Form 6b v2.0
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Functioning Short Form 6b assesses one's ability to engage in physical activities. Raw scores on the survey are converted to T scores, which are standardized scores based on the average in the population; a score of 50 would indicate meeting the average (mean) physical function T score in the reference general population, with a standard deviation of 10. Higher T scores reflect greater physical function and ability to carry out physical activities.
Time Frame: Baseline (0 weeks), Post-test (1 week after intervention completion)
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Experimental: GetActive+
Number analyzed (Participants) | 33
T score
  Baseline | 38.7 (7.3)
  Post-test | 43.2 (8.7)

10. Secondary Outcome: The Interpersonal Support Evaluation List (ISEL-12),
Description: The Interpersonal Support Evaluation List (ISEL-12) measures perceptions of social support. Minimum = 12, Maximum = 48. Higher scores indicate a better outcome.
Time Frame: Baseline (0 weeks), Post-test (1 week after intervention completion)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental: GetActive+
Number analyzed (Participants) | 33
units on a scale
  Baseline | 35.4 (7.8)
  Post-test | 36.5 (7.1)

11. Secondary Outcome: Pain Catastrophizing Scale (PCS)
Description: The Pain Catastrophizing Scale (PCS) is a 13-item measure that assesses hopelessness, helplessness and rumination about pain. Subscales (rumination, magnification, and helplessness) are calculated by summing item responses for the associated questions, and then combined (summed) to create the total score. Items range from 0-4, and total scores range from 0-52. For the subscales, rumination ranges from 0-16, magnification ranges from 0-12, and helplessness ranges from 0-24. Higher scores (on subscales and the scale as a whole) indicate higher levels of pain catastrophizing, i.e. higher scores indicate poorer outcomes. Both subscales and total score are shown here. The means reported reflect the mean of each subscale or total score among GetActive+ participants at the indicated timepoint.
Time Frame: Baseline (0 weeks), Post-test (1 week after intervention completion)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: GetActive+
Number analyzed (Participants) | 33
score on a scale
  Total Score - Baseline | 20.6 (14.5)
  Total score - Post-test | 15.5 (11.4)
  Rumination- Baseline | 7.3 (5.0)
  Rumination- Post-test | 5.7 (4.1)
  Magnification - Baseline | 4.2 (3.8)
  Magnification - Post-test | 3.3 (2.7)
  Helplessness - Baseline | 9.1 (6.7)
  Helplessness - Post-test | 6.6 (5.4)

12. Secondary Outcome: Pain, Enjoyment of Life and General Activity Scale (PEG)
Description: The Pain, Enjoyment of Life and General Activity scale (PEG) rates a participant's pain intensity and related interference in enjoyment of life and general activity. Items are scored on a scale of 0-10, with 0 being no pain (or interference) and 10 being pain as bad as you can imagine (or complete interference). The total score is a sum of the three individual items (Pain Intensity Average, Activity Interference, Enjoyment Interference) divided by 3, with a minimum possible score of 0 and a maximum possible score of 10. Higher scores indicate worse outcomes (i.e. more pain intensity and interference). Scores presented here are the mean total score and mean item scores at the indicated timepoints.
Time Frame: Baseline (0 weeks), Post-test (1 week after intervention completion)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: GetActive+
Number analyzed (Participants) | 33
score on a scale
  Total Score (Baseline) | 6.0 (2.2)
  Total Score (Posttest) | 4.6 (2.6)
  Average Pain Intensity (Baseline) | 6.5 (1.8)
  Average Pain Intensity (Posttest) | 5.4 (2.4)
  Activity Interference (Baseline) | 5.5 (2.9)
  Activity Interference (Posttest) | 4.1 (3.0)
  Enjoyment Interference (Baseline) | 5.8 (2.7)
  Enjoyment Interference (Posttest) | 3.8 (3.0)

13. Secondary Outcome: Applied Mindfulness Process Scale (AMPS)
Description: The Applied Mindfulness Process Scale (AMPS) assesses how participants use mindfulness when facing challenges in daily life. Sum all 15 items to obtain a total score ranging from 0-60. Higher scores indicate higher utilization of mindfulness
Time Frame: Baseline (0 weeks), Post-test (1 week after intervention completion)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental: GetActive+
Number analyzed (Participants) | 33
units on a scale
  Baseline | 37.4 (12.9)
  Post-test | 43.0 (9.7)

14. Secondary Outcome: Cognitive and Affective Mindfulness Scale - Revised (CAMS-R)
Description: Cognitive and Affective Mindfulness Scale - Revised (CAMS-R) rates a participant's broad conceptualization of mindfulness,. Minimum = 12 Maximum = 48. Higher values reflect higher levels of mindfulness.
Time Frame: Baseline (0 weeks), Post-test (1 week after intervention completion)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental: GetActive+
Number analyzed (Participants) | 33
units on a scale
  Baseline | 35.3 (7.2)
  Post-test | 36.0 (6.0)

15. Secondary Outcome: Perceived Stress Scale (PSS-4)
Description: The Perceived Stress Scale (PSS-4) assesses stress perception levels. Total sum of scores. Minimum = 0 Maximum =16; Higher scores are correlated to more stress.
Time Frame: Baseline (0 weeks), Post-test (1 week after intervention completion)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental: GetActive+
Number analyzed (Participants) | 33
units on a scale
  Baseline | 6.7 (2.0)
  Post-test | 5.6 (2.7)

16. Secondary Outcome: Post-Traumatic Checklist-Civilian Version-6 (PCL-C Short Form)
Description: The Post-Traumatic Checklist-Civilian Version-6 (PCL-C short form) assesses current Post Traumatic Stress Disorder symptoms. Items in the measure are scored on a scale of 1-5, with 5 indicating being extremely bothered by a problem (related to stressful experiences) in the past month, and 1 indicating not being bothered at all. The total score is a sum of all item responses; this can range from 6 - 30. Higher scores are suggestive of difficulties with post-traumatic stress, and further assessment and possibly referral for treatment may be indicated especially if a score is 14 or more.
Time Frame: Baseline (0 weeks), Post-test (1 week after intervention completion)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental: GetActive+
Number analyzed (Participants) | 33
units on a scale
  Baseline | 12.5 (5.4)
  Post-test | 11.8 (6.0)

17. Secondary Outcome: Pittsburgh Sleep Quality Index (PSQI) - Sleep Duration
Description: The Pittsburgh Sleep Quality Index (PSQI) is a four-question measure assessing sleep quality. This study ONLY utilized question 4 of the measure, which asks about sleep duration in hours and minutes per night (the time spent actually asleep, not just in bed). Reported below as an outcome is the mean hours of sleep reported by participants at baseline and posttest, i.e. the mean hours reported by participants as captured in Question 4 only of the PSQI measure.
Time Frame: Baseline (0 weeks), Post-test (1 week after intervention completion)
Population: 23 participants provided this information at baseline, but only 19 participants provided it at posttest.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | GetActive+
Number analyzed (Participants) | 23
hours
  Baseline | 5.50 (1.98)
  Posttest: number analyzed (Participants) | 19
  Posttest | 6.23 (2.14)

18. Secondary Outcome: PROMIS Sleep Disturbance - Short Form 6a v1.0
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance Short Form 6a v1.0 assesses quality of sleep. Raw scores on the survey are converted to T scores, which are standardized scores based on the average in the population; a score of 50 would indicate meeting the T score for the average quality of sleep in the reference general population, with a standard deviation of 10. Higher T scores reflect greater sleep disturbance, and thus worse outcomes. The means reported are the mean T scores at the indicated timepoint.
Time Frame: Baseline (0 weeks), Post-test (1 week after intervention completion)
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Experimental: GetActive+
Number analyzed (Participants) | 33
T-score
  Baseline | 55.6 (9.3)
  Post-test | 52.2 (9.9)

19. Secondary Outcome: Everyday Discrimination Scale - Short (EDS-S)
Description: The Everyday Discrimination Scale - Short (EDS-S) assesses the frequency of experiences of discrimination. Each item is scored on a scale of 0-5, with 0 indicating never experiencing that situation, and 5 indicating experiencing it almost every day. Responses are then summed across items, with final scores ranging from 0 - 25. Higher scores indicate greater frequency of discriminatory experiences.
Time Frame: Baseline (0 weeks), Post-test (1 week after intervention completion)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental: GetActive+
Number analyzed (Participants) | 33
units on a scale
  Baseline | 2.9 (3.5)
  Post-test | 2.5 (2.9)

20. Secondary Outcome: Tobacco, Alcohol, Prescription Medications, and Other Substance (TAPS)
Description: The Tobacco, Alcohol, Prescription medications, and other Substance (TAPS) assess substance use behaviors. No summary score. Each item is scored individually for each substance. For each item, higher scores indicate better outcome.
Time Frame: Baseline (0 weeks), Post-test (1 week after intervention completion)
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: GetActive+
Number analyzed (Participants) | 33
Participants
  Tobacco Use: Never | 32
  Tobacco Use: Less than monthly | 1
  Tobacco Use: Monthly | 0
  Tobacco Use: Weekly | 0
  Tobacco Use: Daily or almost daily | 0
  Tobacco Use: Prefer not to respond | 0
  Binge Drinking: Never | 23
  Binge Drinking: Less than monthly | 3
  Binge Drinking: Monthly | 4
  Binge Drinking: Weekly | 0
  Binge Drinking: Daily or almost daily | 0
  Binge Drinking: Prefer not to respond | 3
  Prescription Drug Use: Never | 31
  Prescription Drug Use: Less than monthly | 2
  Prescription Drug Use: Monthly | 0
  Prescription Drug Use: Weekly | 0
  Prescription Drug Use: Daily or almost daily | 0
  Prescription Drug Use: Prefer not to respond | 0

21. Secondary Outcome: Contrast Avoidance Questionnaire - Shortened (CAQ-S)
Description: Contrast Avoidance Questionnaire - Shortened (CAQ-S) a measure of sustaining negative emotionality to protect against sudden shifts in emotion. Minimum = 8, Maximum = 40 with higher scores indicating worse outcomes.
Time Frame: Baseline (0 weeks), Post-test (1 week after intervention completion)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental: GetActive+
Number analyzed (Participants) | 33
units on a scale
  Baseline | 13.7 (6.1)
  Post-test | 12.9 (4.9)

22. Secondary Outcome: Patient Global Impression of Change (PGIC)
Description: The Patient Global Impression of Change (PGIC) measures changes in pain in response to treatment. Minimum = 0, Maximum = 6. Higher scores indicate worse outcome.
Time Frame: Baseline (0 weeks), Post-test (1 week after intervention completion)
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: GetActive+
Number analyzed (Participants) | 31
Participants
  Very much improved | 11
  Much improved | 7
  Minimally improved | 6
  No change | 5
  Minimally worse | 2
  Much worse or very much worse | 0

23. Secondary Outcome: Tampa Scale for Kinesiophobia-11 (TSK11)
Description: The Tampa Scale for Kinesiophobia-11 (TSK11) is an 11-item questionnaire that assesses fear avoidance and fear of activity. Summary score of total responses with Minimum = 11 and Maximum = 44. Higher scores indicate higher kinesiophobia.
Time Frame: Baseline (0 weeks), Post-test (1 week after intervention completion)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental: GetActive+
Number analyzed (Participants) | 33
units on a scale
  Baseline | 28.9 (6.7)
  Post-test | 25.5 (5.9)

24. Secondary Outcome: UCLA-3 Loneliness Scale
Description: The UCLA-3 Loneliness Scale measures isolation / perceived lack of social connectedness. Minimum = 3, Maximum = 9. Higher scores indicate worse outcome.
Time Frame: Baseline (0 weeks), Post-test (1 week after intervention completion)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental: GetActive+
Number analyzed (Participants) | 33
units on a scale
  Baseline | 5.1 (2.0)
  Post-test | 4.8 (1.8)

25. Secondary Outcome: Measure of Current Status (MOCS)
Description: The MOCS questionnaire assesses ability to engage in a series of healthy coping skills (e.g., relaxation, social support, adaptive thinking). Minimum = 0, maximum = 52. Higher scores indicate better outcome and a stronger ability to recognize stress and cope.
Time Frame: Baseline (0 weeks), Post-test (1 week after intervention completion)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental: GetActive+
Number analyzed (Participants) | 33
units on a scale
  Baseline | 28.8 (9.8)
  Post-test | 32.0 (9.4)

26. Secondary Outcome: Self-Compassion Scale - Short Form (SCS-SF)
Description: The Self-Compassion Scale - Short Form (SCS-SF) is the rate of a participant's amount of self-compassion. Scores are calculated by averaging the 12 items with Minimum = 1, Maximum = 5. Higher scores indicate worse outcome.
Time Frame: Baseline (0 weeks), Post-test (1 week after intervention completion)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental: GetActive+
Number analyzed (Participants) | 33
units on a scale
  Baseline | 3.4 (0.7)
  Post-test | 3.6 (0.8)

27. Secondary Outcome: Gratitude Questionnaire (GQ-6)
Description: The Gratitude Questionnaire (GQ-6) assesses the proneness to experience gratitude in daily life. All items individual items are scored from 1=strongly disagree to 7=strongly agree. The total score is a sum of all the items, with a minimum of 6 and maximum of 42. Higher scores indicate a greater amount of gratitude. Results are reported for baseline and posttest (timepoint indicated by the row title description)>
Time Frame: Baseline (0 weeks), Post-test (1 week after intervention completion)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GetActive+
Number analyzed (Participants) | 32
score on a scale
  Baseline | 35.00 (5.66)
  Posttest | 35.13 (5.73)

28. Other Pre Specified Outcome: Qualitative Assessment of Intervention by Participants
Description: Qualitative information was collected from patients through one-on-one exit interviews assessing perceptions of intervention; these were completely qualitative (i.e. held through discussions and not by using surveys or structured questions, etc). The reported result is the number of participants who completed this optional exit interview after intervention completion.
Time Frame: Post-test (1 week after intervention completion)
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: GetActive+
Number analyzed (Participants) | 33
Participants | 32

ADVERSE EVENTS:
Time Frame: Adverse events were monitored for each participant over the course of their participation in the intervention (10 weeks) through posttest (which was 1 week after the intervention was completed). The total counts of adverse events reported here reflect the total counts of all the events of all study participants, taken over the duration of the study (which was 11 months long in total)
Arm/Group | Experimental: GetActive+
All-Cause Mortality (participants affected / at risk) | 0/33
Serious Adverse Events (participants affected / at risk) | 3/33
Other Adverse Events (participants affected / at risk) | 17/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: GetActive+ (N=33)
Kidney Stones and Infection (General disorders) | 1 (1) — Hospitalization due to kidney stone surgery and consequent infection.
Suicide attempt, Command hallucinations for suicide (Psychiatric disorders) | 1 (1) — Report of suicide attempt and hearing near constant thoughts of suicide.
Adverse effect of drug or medicament (Injury, poisoning and procedural complications) | 1 (1) — Hospitalization due to complications from new medication.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: GetActive+ (N=33)
Musculoskeletal pain/injury (Musculoskeletal and connective tissue disorders) | 4 (6)
Fall on same level from slipping, tripping or stumbling (Musculoskeletal and connective tissue disorders) | 5 (5)
Severe Nosebleed (Epistaxis) (Blood and lymphatic system disorders) | 1 (1)
Kidney Stones (Renal and urinary disorders) | 1 (1)
Syncopal Episode (Nervous system disorders) | 1 (1)
Fall on or from stairs or steps (Musculoskeletal and connective tissue disorders) | 2 (2)
Thrombophlebitis (Cardiac disorders) | 1 (1)
Arrhythmias (Cardiac disorders) | 2 (3) — One arrhythmia episode was accompanied by dizziness and temporary hearing loss in right ear.
Fall from furniture (Musculoskeletal and connective tissue disorders) | 1 (1)
Diverticulitis (Gastrointestinal disorders) | 1 (1)
Concern regarding prior hip replacement (Surgical and medical procedures) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-04-16): https://cdn.clinicaltrials.gov/large-docs/31/NCT05782231/Prot_SAP_000.pdf
  • Informed Consent Form (2023-07-31): https://cdn.clinicaltrials.gov/large-docs/31/NCT05782231/ICF_001.pdf